CLINICAL TRIAL: NCT02431169
Title: Genomic Landscape of EGFR Mutant NSCLC Prior to Erlotinib and at the Time of Disease Progression Following Erlotinib
Brief Title: Genomic Landscape of EGFR Mutant NSCLC Prior to Erlotinib and at the Time of Disease Progression
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201407158
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Carcinoma, Non-Small-Cell-Lung; Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Specimen (tissue and blood) acquisition will take place under Washington University's study HRPO# 201305031 and will be analyzed under this study.
  * Fresh tissue will be taken at the time of diagnosis of metastatic disease and again at progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose to conduct a pilot feasibility study of single agent erlotinib in patients with metastatic EGFR mutant adenocarcinoma of the lung with up to one prior treatment with the sole purpose of characterizing the genomic landscape before erlotinib and at the time of disease progression. The logistics of obtaining adequate quality fresh tissue specimens for sequencing studies before therapy and at the time of disease progression in patients with advanced lung cancer are complex and a thorough understanding of the practical challenges in conducting a study like this is crucial.

The current proposal will include exome and transcriptome sequencing from blood collected at baseline along with tumor samples obtained prior to starting erlotinib and at the time of disease progression (a total of two tissue samples and one blood sample per patient). If carried out successfully, the proposed strategy very likely will lead to a larger and adequately powered study to understand fully evolving molecular changes due to clonal selection under treatment pressure. The pace of progress in the field of sequencing technology currently underway is only likely to accelerate in the near future yielding richer and highly content-rich information. Moreover, it is likely that genomic information from DNA sequencing and transcriptome will be supplemented by analyses of translatomes and proteomes.

The investigators plan to sequence paired tumor specimens from 20 patients with EGFR mutant adenocarcinoma of the lung before treatment with erlotinib and at the time of disease progression following treatment with erlotinib. As the investigators expect some drop off (due to unexpected clinical events precluding a second biopsy at the time of disease progression, poor specimen quality and early discontinuation of therapy for non-progression), the investigators will enroll 40 patients in this trial to get 20-paired specimens.

ELIGIBILITY:
Patient Selection

* Diagnosis of metastatic stage IIIB/IV lung adenocarcinoma
* Presence of known sensitizing mutations in EGFR TK domain
* Consented to HRPO# 201305031 ("Tissue and Blood Acquisition for Genomic Analysis and Collection of Health Information from Patients with Thoracic Malignancies, Suspected -Thoracic Malignancies, or Mesothelioma")
* Treatment with standard of care erlotinib
* At least 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of participants with stage IIIB/IV non-small cell lung cancer with presence of known sensitizing mutations in the EGFR TK domain and absense of known resistant mutations in the EGFT TK domain.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Genetic changes associated with disease progression following treatment with erlotinib in patients with activating mutations in the EGFR TK domain known to be responsive to therapy | Up to 3 years
  Exome and transcriptome sequencing of tumor before therapy with erlotinib and at the time of relapse. In addition, exome sequencing of peripheral blood DNA will be done (for germ line).

SECONDARY OUTCOMES:
Correlate mutations in signaling kinases with therapeutic response | Up to 3 years
Correlate the allelic ratio of wild type to mutant EGFR with duration of response | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu